CLINICAL TRIAL: NCT02202499
Title: Translating Extinction Research to Improve Pharmacotherapy for Tobacco Dependence: Intervention Development and Feasibility Trial
Brief Title: Translating Extinction Research to Improve Pharmacotherapy for Tobacco Dependence
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: James and Esther King Biomedical Research Program (Other); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MCC-17654
Record Dates: First submitted 2014-07-22; First posted 2014-07-29 (Estimated); Results first posted 2019-07-25 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Smoking Cessation; Tobacco Dependence
Keywords: pharmacotherapy
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder | interventions — Varenicline; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Extended Varenicline + Facilitated Extinction (Active Comparator): Extended Varenicline plus Facilitated Extinction (EV+FE). Participants in the EV+FE condition will receive varenicline for a 4-week run-in period while continuing to smoke. In addition, the EV+FE condition will receive counseling and support materials (including a review and self-monitoring workbook tentatively titled, Winding Down: A Guide to Quitting Smoking using Varenicline) instructing participants to systematically utilize the FE techniques provided. All groups will undergo periodic laboratory assessments and surveys.
  Interventions: Drug: Varenicline; Other: Counseling and Support Materials; Other: Laboratory Assessments
- Standard Varenicline (SV) (Active Comparator): Participants in the Standard Varenicline (SV) condition will receive varenicline for the usual 1-week run-in period while continuing to smoke. All groups will undergo periodic laboratory assessments and surveys.
  Interventions: Drug: Varenicline; Other: Laboratory Assessments
- Extended Varenicline (EV) (Active Comparator): Participants in the Extended Varenicline (EV) condition will receive varenicline for a 4-week run-in period while continuing to smoke. All groups will undergo periodic laboratory assessments and surveys.
  Interventions: Drug: Varenicline; Other: Laboratory Assessments

INTERVENTIONS:
Drug: Varenicline — All participants will take the following dose of varenicline: 0.5 mg once a day on days 1-3, 0.5 mg twice a day on days 4-7, and 1 mg twice a day through week 16 of the study. Arm descriptions show specific details for each group.
  Other Names: Chantix™
Other: Counseling and Support Materials — Counseling and support materials (including a review and self-monitoring workbook tentatively titled, Winding Down: A Guide to Quitting Smoking using Varenicline) instructing participants to systematically utilize the FE techniques provided.
  Arms: Extended Varenicline + Facilitated Extinction
Other: Laboratory Assessments — The first laboratory assessment will consist of completion of questionnaires and a cue-reactivity test. The second laboratory assessment will be scheduled for the end of the week before the participant's quit date. It will involve completion of questionnaires and another cue reactivity test. A follow-up session conducted by research staff will occur one month after the target quit date to collect information about each participant's current smoking status, smoking rate, varenicline use, and opinion about the treatment. A second follow-up session will be conducted by telephone and will occur three months after the target quit date, at the end of varenicline use. At the end of the study, participants will be asked to complete a brief survey asking basic information, similar to the questions during the screening period.

SUMMARY:
The purpose of this Pilot feasibility study is to find out the effect of different behavioral treatments along with different duration of a drug called varenicline, on smoking behavior and quitting smoking. Varenicline, also known as Chantix™, is an FDA-approved medication that has been shown to help people quit smoking.

DETAILED DESCRIPTION:
Following the initial telephone screening, eligible participants will be scheduled for a screening evaluation session.

Following the screening evaluation, participants who pass the medical screening and meet all other inclusion criteria will be scheduled for their first assessment and then randomized to receive standard varenicline (SV), extended varenicline (EV), or extended varenicline plus facilitated extinction (EV + FE). The randomization list will be generated by the study statistician. It will be stratified by gender and will employ a variable block randomization that will guarantee that the arms are balanced when a given block is filled.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Smoke at least 10 cigarettes daily for the past year
* Expired-air carbon monoxide (CO) > 8 ppm
* Medically eligible to receive varenicline
* Score at least a 5 on the Contemplation Ladder (Biener & Abrams 1991), a measure of motivation to quit smoking.

Exclusion Criteria:

* Are pregnant or lactating
* Have renal dysfunction
* Have a history of seizures
* Are medically at risk in the judgment of the study physician
* Have ever used varenicline
* Have used other smoking cessation medications within the past three months
* Have current psychiatric disorders (i.e. major depression, bipolar, and/or psychotic disorders)
* Have substance use disorder as determined by a psychiatric screener (Mini International Neuropsychiatric Interview [MINI]; Sheehan et al 2015).
* We must limit the number of participants from the same street address to 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2014-07-17 (Actual); Primary Completion 2015-12-11 (Actual); Study Completion 2019-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Brandon, Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Daily cigarette smokers were recruited from the community for a smoking cessation intervention study, from July 2014 through August 2015, by Moffitt Cancer Center in Tampa, Florida.
Pre-assignment Details: 86 interested parties were consented, 1 later declined, 23 did not meet criteria. 62 were eligible, 3 discontinued due to factors unrelated to study, 1 failed to attend first assessment. 58 parties participated in the study.
Groups:
- Extended Varenicline + Facilitated Extinction: Active Comparator: Extended Varenicline + Facilitated Extinction.
- Standard Varenicline: Active Comparator: Standard Varenicline (SV).
- Extended Varenicline: Active Comparator: Extended Varenicline (EV).
Period: Overall Study
Arm/Group | Extended Varenicline + Facilitated Extinction | Standard Varenicline | Extended Varenicline
Started | 21 | 20 | 21
Completed | 19 | 20 | 19
Not Completed | 2 | 0 | 2
Not completed — Cancer diagnosis | 0 | 0 | 1
Not completed — Moved from area | 0 | 0 | 1
Not completed — Declined before randomization | 1 | 0 | 0
Not completed — Auto accident | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Extended Varenicline + Facilitated Extinction | Standard Varenicline | Extended Varenicline | Total
Number analyzed (Participants) | 19 | 20 | 19 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (50.5) | 51.9 (11.0) | 48.4 (11.4) | 50.5 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 9 | 25
  Male | 12 | 11 | 10 | 33
Region of Enrollment [Number; unit: participants]
  United States | 19 | 20 | 19 | 58

OUTCOME MEASURES:

1. Primary Outcome: Rate of Participant Retention
Description: Practicality: Number of participants completing 3 month post treatment follow-up. Feasibility: Ability to recruit and retain sufficient numbers of the target population, which would be essential in conducting a future randomized clinical trial (RCT).
Time Frame: End of post treatment follow-up period of 3 months - approximately 28 weeks
Population: All participants who completed 3 month post treatment follow up, regardless of study arm
Measure: Count of Participants; unit: Participants
Groups:
- Extended Varenicline + Facilitated Extinction: All participants who received Extended Varenicline + Facilitated Extinction
- Standard Vareniclline: All participants who received Standard Varenicline (SV)
- Extended Varenicline: All participants who received Extended Varenicline
Arm/Group | Extended Varenicline + Facilitated Extinction | Standard Vareniclline | Extended Varenicline
Number analyzed (Participants) | 19 | 20 | 19
Participants | 15 | 16 | 19

2. Secondary Outcome: Client Satisfaction Questionnaire (CSQ) Results
Description: Acceptability: Mean score of Client Satisfaction Questionnaire (CSQ) version 8 by Attkison & Greenfield. Questionnaire scores client satisfaction with a scale of 1-4 per question, 1 being very dissatisfied and 4 being very satisfied. Score total range is 8-32. A total score of 32 would be the highest possible Client Satisfaction Score.
Time Frame: One month post treatment - approximately 20 weeks
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Extended Varenicline + Facilitated Extinction: All participants who received Extended Varenicline +Facilitated Extinction
- Standard Vareniclline: All participants who received Standard Varenicline
Arm/Group | Extended Varenicline + Facilitated Extinction | Standard Vareniclline | Extended Varenicline
Number analyzed (Participants) | 19 | 20 | 19
units on a scale | 30.33 [23 to 32] | 30.80 [27 to 32] | 30.47 [25 to 32]

3. Secondary Outcome: Rate of Intervention Adherence - Medication
Description: Percent of participants still using varenicline at time of analysis.
Time Frame: One month post treatment - approximately 20 weeks
Population: All participants.
Measure: Number; unit: percentage of participants
Arm/Group | Extended Varenicline + Facilitated Extinction | Standard Varenicline | Extended Varenicline
Number analyzed (Participants) | 19 | 20 | 19
percentage of participants | 80 | 80 | 84

4. Secondary Outcome: Average Intervention Adherence - Cigarettes Per Day (CPD)
Description: Average Cigarettes per Day across group, during last week of treatment.
Time Frame: During last week of treatment, week 16
Population: All participants.
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | Extended Varenicline + Facilitated Extinction | Standard Varenicline | Extended Varenicline
Number analyzed (Participants) | 19 | 20 | 19
cigarettes per day | 17.58 (5.85) | 14.95 (9.06) | 11.05 (6.16)

5. Secondary Outcome: Mean Peak Craving Score Per Group
Description: Peak craving per day by treatment group, scored using an 11-point Likert scale 0-10. 0 was "none", 5 "medium" and 10 "very high/strong"
Time Frame: Across 4 pre-quit weeks
Population: All participants.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Extended Varenicline + Facilitated Extinction | Standard Varenicline | Extended Varenicline
Number analyzed (Participants) | 19 | 20 | 19
units on a scale | 4.64 (0.56) | 6.34 (0.49) | 4.56 (0.34)

6. Secondary Outcome: Mean Smoking Satisfaction Score Per Group
Description: Smoking satisfaction per day by treatment group, using 11-point Likert scale, 0-10. 0 was "none", 5 "medium" and 10 "very high"
Time Frame: Across 4 pre-quit weeks
Population: All participants.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Extended Varenicline + Facilitated Extinction | Standard Varenicline | Extended Varenicline
Number analyzed (Participants) | 19 | 20 | 19
units on a scale | 3.37 (0.64) | 5.22 (067) | 2.59 (0.40)

ADVERSE EVENTS:
Time Frame: 15 weeks
Description: Adverse Events collected after start of Varenicline until end of treatment (15 weeks)
Arm/Group | Extended Varenicline + Facilitated Extinction | Standard Varenicline | Extended Varenicline
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 1/19 | 1/20 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/20 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extended Varenicline + Facilitated Extinction (N=19) | Standard Varenicline (N=20) | Extended Varenicline (N=19)
Cardiac Disorders - Other (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Esophageal Ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gallblader Pain (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint range of motion decreased lumbar spine (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes